CLINICAL TRIAL: NCT03877276
Title: Dietary Oxalate and Immune Cell Function
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Tanecia Mitchell, PhD, Principal Investigator, University of Alabama at Birmingham
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: F151123009
Record Dates: First submitted 2019-03-05; First posted 2019-03-15 (Actual); Last update posted 2025-06-09 (Actual); Status verified 2025-06

CONDITIONS: Kidney Stone
Keywords: dietary oxalate; diet therapy
MeSH Terms: conditions — Kidney Calculi | interventions — Breakfast

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (8):
- 3d Diet+Spinach Smoothie+Breakfast (Experimental): 3 days of prepared meals with fasting on the final day. On final day, participants will return to study site and drink a prepared blended spinach smoothie and be provided a breakfast meal.
  Interventions: Dietary Supplement: Breakfast; Dietary Supplement: Spinach smoothie
- 5d Diet+Spinach Smoothie+Breakfast (Experimental): 5 days of prepared meals with fasting on the final day. On final day, participants will return to the study site and drink a prepared blended spinach smoothie and be provided a breakfast meal.
  Interventions: Dietary Supplement: Breakfast; Dietary Supplement: Spinach smoothie
- 3d Diet+Kale Smoothie+Breakfast (Experimental): 3 days of prepared meals with fasting on the final day. On the final day, participants will return to the study site and drink a prepared kale smoothie and be provided a breakfast meal.
  Interventions: Dietary Supplement: Breakfast; Dietary Supplement: Kale smoothie
- 3d Diet+V Spinach Smoothie+Breakfast (Experimental): 3 days of prepared meals with fasting on the final day. On final day, participants will return to the study site and drink a prepared blended spinach smoothie with varying amounts of spinach and be provided a breakfast meal.
  Interventions: Dietary Supplement: Breakfast; Dietary Supplement: V spinach smoothie
- 3d Diet+Blended Smoothie+Breakfast (Experimental): 3 days of prepared meals with fasting on the final day. On final day, participants will return to the study site and drink a prepared blended smoothie and be provided a breakfast meal.
  Interventions: Dietary Supplement: Breakfast; Dietary Supplement: Blended smoothie
- 3d Diet+Breakfast (Experimental): 3 days of prepared meals with fasting on the final day. On final day, participants will return to the study site and be provided a breakfast meal.
  Interventions: Dietary Supplement: Breakfast
- 3d Diet+Sodium Oxalate Drink+Breakfast (Experimental): 3 days of prepared meals with fasting on the final day. On final day, participants will return to the study site and drink a prepared sodium oxalate drink and be provided a breakfast meal.
  Interventions: Dietary Supplement: Breakfast; Dietary Supplement: Sodium oxalate drink
- 3d Diet+Spinach Smoothie+Breakfast w/ 24 Hr Urine (Experimental): 3 days of prepared meals with fasting on the final day. On final day, participants will return to the study site and drink a blended spinach smoothie and be provided a breakfast meal.
  Interventions: Dietary Supplement: Breakfast; Dietary Supplement: Spinach smoothie

INTERVENTIONS:
Dietary Supplement: Breakfast — a prepared meal consisting of pastry and 2 cooked egg whites
Dietary Supplement: Spinach smoothie — a prepared blended spinach smoothie, consisting of banana, avocado, orange juice, and spinach
  Arms: 3d Diet+Spinach Smoothie+Breakfast; 3d Diet+Spinach Smoothie+Breakfast w/ 24 Hr Urine; 5d Diet+Spinach Smoothie+Breakfast
Dietary Supplement: Kale smoothie — prepared blended kale smoothie, consisting of banana, avocado, orange juice, and kale
  Arms: 3d Diet+Kale Smoothie+Breakfast
Dietary Supplement: Blended smoothie — a prepared blended smoothie, consisting of banana, avocado, and orange juice
  Arms: 3d Diet+Blended Smoothie+Breakfast
Dietary Supplement: V spinach smoothie — a prepared blended spinach smoothie, consisting of banana, avocado, orange juice, and a varying amount (low, medium, high) of spinach
  Arms: 3d Diet+V Spinach Smoothie+Breakfast
Dietary Supplement: Sodium oxalate drink — a prepared sodium oxalate drink
  Arms: 3d Diet+Sodium Oxalate Drink+Breakfast

SUMMARY:
The purpose of this study is to evaluate mitochondrial function in white blood cells and platelets from healthy individuals following dietary oxalate intake.

DETAILED DESCRIPTION:
Inflammation and dietary oxalate have been shown to play an important role in the development of kidney stones. Oxalate is a small molecule found in plants and plant-derived food. Individuals that have high oxalate intake have an increased risk of developing kidney stones. The co-investigators have previously shown that healthy subjects that consume dietary oxalate have increased plasma and urine oxalate.

White blood cells are essential for the immune response and rely on the mitochondria to carry out important cell functions. The Principal Investigator's current research shows that patients with calcium oxalate kidney stones have decreased mitochondrial function in their immune cells. Using the expertise of the investigators, this study will test whether oxalate has a direct effect on mitochondrial function in immune cells from healthy subjects. This information could help us understand the role of oxalate on the immune system during kidney stone pathogenesis.

ELIGIBILITY:
Inclusion Criteria:

* Mentally competent adults who are able to read and comprehend the consent form, written in English
* Male or Female
* Age 18 to 70 years
* Non-tobacco users
* BMI between 19 and 27
* Willingness to abstain from vigorous exercise during study period
* Normal blood comprehensive metabolic panel

Exclusion Criteria:

* Mentally incompetent adults who are unable to read or comprehend the consent form, written in English
* Pregnant females
* Active medical problems
* History of kidney stones
* Any medical disorder that could influence absorption or excretion of oxalate
* BMI less than 19 or greater than 27
* Tobacco users
* Current use of medications or dietary supplements

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2016-07-21 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in monocyte cellular energetics after 5 hours | 0 hours - 5 hours
  Cellular bioenergetics (oxygen consumption rate) will be measured in isolated monocytes from human blood using a Seahorse XF Analyzer machine. Monocyte cellular bioenergetics will be measured before and after consuming a spinach smoothie (pre- and post-loads; Time 0 hours and 5 hours) to assess a change in monocyte cellular energetics after 5 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Tanecia Mitchell, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kumar P, Patel M, Oster RA, Yarlagadda V, Ambrosetti A, Assimos DG, Mitchell T. Dietary Oxalate Loading Impacts Monocyte Metabolism and Inflammatory Signaling in Humans. Front Immunol. 2021 Feb 25;12:617508. doi: 10.3389/fimmu.2021.617508. eCollection 2021. PMID 33732242